CLINICAL TRIAL: NCT00371202
Title: Comparison of Penetrating Keratoplasty and Deep Lamellar Keratoplasty With the Big Bubble Technique for Keratoconus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8390
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2007-01

CONDITIONS: Keratoconus
Keywords: keratoconus, penetrating keratoplasty,; deep lamellar keratoplasty; big bubble technique
MeSH Terms: conditions — Keratoconus | interventions — Corneal Transplantation

INTERVENTIONS:
Procedure: keratoplasty

SUMMARY:
it is a randomized clinical trial to compare deep lamellar keratoplasty (DLK) Using big bubble technique and Penetrating Keratoplasty (PK) in patients with keratoconus

DETAILED DESCRIPTION:
In this randomized clinical trial 50 keratoconic eyes of 50 patients randomly assigned in two groups: 25 patients underwent DLK with the big bubble technique and the other 25 patients underwent PK with the standard technique using hessburg - Barron trephine. One surgeon performed all operations using a 16 bites separate 10-0 nylon sutures. We used A-scan ultrasonic biometry for measuring vitreous length (VL) before surgery. If VL≥15.50mm, a trephine 0.25mm larger than recipient and if VL was <15.50mm, a trephine 0.50 mm larger than recipient were considered. Selective suture removal was started 3 months after operation. quality of vision endothelial cell changes and correlation between refractive outcome and VL in relation to donor-recipient disparity, were measured and analyzed in both PK and DLK 15 mos postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe keratoconus
* contact lens intolerance
* low visual acuity due to anterior stromal scar
* age between 15 to 50 years

Exclusion Criteria:

* posterior stromal scar with descemets membrane involvement
* history of hydrops
* fuchs endothelial dystrophy
* glaucoma
* cataract
* history of intraocular surgery
* history of vernal keratoconjunctivitis
* intraoperative complications
* reoperation (resuturing- regraft)

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2006-07; Study Completion 2006-08

PRIMARY OUTCOMES:
Uncorrected visual acuity (UCVA), best corrected visual acuity(bcva), refractive astigmatism, endothelial cell density, mean cell area, polymegathism (CV), Contrast sensitivity, Root-mean-square (RMS) Wavefront error, Pearson correlation factor between

CONTACTS AND LOCATIONS:
Overall Officials: Bahram Einollahi, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Bahram Einollhi, MD, Tehran, Tehran Province, Iran